CLINICAL TRIAL: NCT01133457
Title: Comparative,Randomized,Single-dose,2-way Crossover Bioavailability Study of Dr.Reddy's Laboratories Limited Finasteride Tablets 1 mg and Merck & Co., Propecia in Healthy Adult Males Under Fed Condition.
Brief Title: Bioequivalence Study of Dr.Reddy's Laboratories Limited Finasteride Tablets 1 mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sr. Manager-Research and Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 012744
Record Dates: First submitted 2010-05-27; First posted 2010-05-28 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2002-03

CONDITIONS: Healthy
Keywords: Bioequivalence,Finasteride,Crossover
MeSH Terms: interventions — Finasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Finasteride (Experimental): Finasteride tablets 1 mg of Dr. Reddy's
  Interventions: Drug: Finasteride
- Propecia (Active Comparator): Propecia 1 mgTablets of Merck & Co.,
  Interventions: Drug: Finasteride

INTERVENTIONS:
Drug: Finasteride — Finasteride tablets 1 mg
  Other Names: Propecia

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Dr. Reddy's Laboratories, Ltd. and Merck & Co. (Propecia®)

1 mg finasteride tablets under fed conditions following administration of a 3 mg dose.

DETAILED DESCRIPTION:
Detailed Description : The study was conducted as an open-label, randomized, single-dose, 2-way crossover, relative bioavailability study performed on 24 healthy adult male volunteers and 2 alternates. A total of 24 subjects completed the clinical phase of the study. In each period, subjects were housed from the evening before dosing until after the 36-hour blood draw. Single oral 3 mg doses were separated by a washout period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

History or presence of significant:

• cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.

In addition, history or presence of:

* alcoholism or drug abuse within the past year;
* hypersensitivity or idiosyncratic reaction to finasteride or any other 5-a reductase inhibitor.

Subjects who have been on an abnormal diet (for whatever reason) during the 28 days preceding the study.

Subjects who, through completion of the study, would have donated in excess of:

* 500 mL of blood in 14 days, or
* 500 - 750 mL of blood in 14 days (unless approved by the Principal Investigator),
* 1000 mL of blood in 90 days,
* 1250 mL of blood in 120 days,
* 1500 mL of blood in 180 days,
* 2000 mL of blood in 270 days,
* 2500 mL of blood in 1 year. Subjects who have participated in another clinical trial within 28 days prior to the first dosing.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-04; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Cohen Street, Saint-laurent, Montreal (quebec), Canada